CLINICAL TRIAL: NCT04443478
Title: Laparoscopic Versus Open Lower Mediastinal Lymphadenectomy for Siewert Type II/III Adenocarcinoma of Esophagogastric Junction: an Exploratory, Prospective, Observational, IDEAL Stage 2, Cohort Study
Brief Title: Laparoscopic Versus Open Lower Mediastinal Lymphadenectomy for Esophagogastric Junction Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Changzhi People's Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Fujian Medical University Union Hospital (Other); Shanghai Zhongshan Hospital (Other); Fudan University (Other); Guangdong Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Hebei Medical University Fourth Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Nanfang Hospital, Southern Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Affiliated Hospital of Qinghai University (Other); The First Affiliated Hospital of Xiamen University (Other); Shandong Provincial Hospital (Other Government); Shanxi Province Cancer Hospital (Other); RenJi Hospital (Other); Ruijin Hospital (Other); Beijing Friendship Hospital (Other); West China Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Zhejiang Cancer Hospital (Other); Chinese PLA General Hospital (Other); First Hospital of China Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, President of Beijing Cancer Hospital, Peking University
Other Study IDs: CLASS-10
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer
Keywords: esophagogastric junction; lower mediastinal lymphadenectomy; laparoscopic gastrectomy; IDEAL framework
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic Surgery: Lower Mediastinal Lymphadenectomy should be finished via laparoscopic method.
  Interventions: Procedure: Radical gastrectomy with dissection of lower mediastinal lymph node
- Open Surgery: Lower Mediastinal Lymphadenectomy should be finished via open method.
  Interventions: Procedure: Radical gastrectomy with dissection of lower mediastinal lymph node

INTERVENTIONS:
Procedure: Radical gastrectomy with dissection of lower mediastinal lymph node — Radical gastrectomy for gastric cancer should be consistent with Japanese gastric cancer treatment guideline.

SUMMARY:
Mediastinal lymph node dissection has been adopted as standard treatment for adenocarcinoma of esophagogastric junction(AEJ). This multi-center, exploratory, prospective, cohort study aims at provide standard technical details of laparoscopic mediastinal lymph node dissection, and explore the potential clinical effects, gather key information for following study regarding sample size calculation, primary outcome and feasibility.

DETAILED DESCRIPTION:
Introduction: Lower mediastinal lymph node dissection has been adopted as standard by treatment guideline for adenocarcinoma of esophagogastric junction(AEJ), but the effect of laparoscopic mediastinal lymph node dissection remains unknown. The aim of this study is to provide standard technical details of laparoscopic mediastinal lymph node dissection, and explore the potential clinical effects, gather key information for following study regarding sample size calculation, primary outcome and feasibility. This study report intervention development, governance procedures and selection and reporting of outcomes to optimize methods for using the Idea, Development, Exploration, Assessment, Long-term follow-up (IDEAL) framework for surgical innovation that informs evidence-based practice.

Methods and analysis: This is an IDEAL stage II, prospective, parallel control, open label, multi-center and exploratory study. The inclusion criteria is Siewert II/ III, AEJ, cT2-4aN0-3M0(AJCC-8th Gastric Cancer TNM stage manual), decide to receive radical gastrectomy, without preoperative anti-neoplastic therapy. The individual included in the study is performed the radical total or proximal gastrectomy plus the lower mediastinal lymphadenectomy via either laparoscopic (trial arm) or open (control arm) TH approach. The surgical approach is determined by the investigator in each center before the operation and recorded in the electronic case report forms (CRF).

The primary outcome is the number of lower mediastinal lymph nodes retrieved. Secondary outcome include complication, surgery length, postoperative death, R0 resection rate, etc. Expected sample size is 518 in each group, thus has 80% power to detect a difference of 0.17 in the average number of lower mediastinal lymph node dissected in between two groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* Karnofsky score ≥70%;Or ECOG score ≤2;
* Preoperative pathological biopsy confirmed adenocarcinoma.
* According to gastroscopy, abdominal CT or upper gastrointestinal angiography, the tumor site conforms to the definition of esophageal and gastric junction adenocarcinoma in the "Chinese expert consensus", that is, the tumor center is within 5cm above and below the esophagogastric anatomical junction and crosses or touches the esophagogastric junction;
* Length of esophageal invasion ≤2cm;
* By abdominal contrast-enhanced CT/MRI, the clinical stage was CT2-4aN0-3M0 (according to AJCC-8th TNM tumor stage);
* Subject's blood routine and biochemical indicators meet the following standards: hemoglobin ≥80g/L; Absolute count of neutrophils (ANC) ≥1.5×109/L; Platelet ≥75×109/L;ALT and AST≤2.5 times the normal upper limit; ALP≤2.5 times the normal upper limit; Serum total bilirubin ≤1.5 times the normal upper limit; Serum creatinine ≤ the normal upper limit; Serum albumin ≥30g/L;
* Obtain written informed consent.

Exclusion Criteria:

* Any anti-cancerous treatment received prior to surgery.
* Multiple malignant lesions in the stomach.
* Suspicious lymph node metastasis in the middle and/or upper mediastinum.
* Surgical history in the upper abdomen (laparoscopic cholecystectomy excluded).
* Pregnant or breastfeeding women.
* Uncontrolled epilepsy, central nervous system disease or mental disorder.
* The Bulky N2 status.
* The emergency surgery.
* Severe heart disease.
* History of cerebral infarction or cerebral hemorrhage within 6 months.
* Organ transplant recipients who need immunosuppressive therapies.
* Other malignancy diagnosed within 5 years (cured dermoid caner and cervical cancer excluded).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically Confirmed esophageal gastric adenocarcinoma, clinical stage cT2-4aN3M0(AJCC - 8th gastric cancer tumor TNM staging), Siewert Ⅱ/Ⅲ, receive surgical treatment without preoperative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1036 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of lower mediastinal lymph nodes retrieved | immediately after the pathology report issued
  The number of lower mediastinal lymph nodes retrieved

SECONDARY OUTCOMES:
Rate of complication during Lower Mediastinal Lymphadenectomy | immediately after the surgery
  Complication during Lower Mediastinal Lymphadenectomy & anastomosis, including damage of pericardium, esophagus, etc.
Rate of postoperative complication after Lower Mediastinal Lymphadenectomy | Day 30 after surgery
  Postoperative complication after Lower Mediastinal Lymphadenectomy, including leakage, bleeding, etc, complication related with Lower Mediastinal Lymphadenectomy
Time length of Lower Mediastinal Lymphadenectomy | immediately after the surgery
  Time length of Lower Mediastinal Lymphadenectomy
Rate of Postoperative complication | Day 30 after surgery
  Any complication within 30d after surgery
Rate of postoperative death | Day 30 after surgery
  death within 30 days after surgery
Rate of unscheduled reoperation | Day 30 after surgery
  reoperation within 30 days after surgery
Rate of unscheduled readmission | Day 30 after surgery
  unscheduled readmission within 30 days after surgery
R0 resection rate | immediately after the pathology report issued
  R0 resection rate
Proximal margin length | 30minutes after removal of tumor
  from proximal tumor margin to proximal margin
Local recurrence of lower mediastinal area in 3 years | Year 3 after surgery
  Local recurrence of lower mediastinal area in 3 years
Rate of cancer specific death in 3 years | Year 3 after surgery
  Rate of cancer specific death in 3 years
Recurrence free survival in 3 years | Year 3 after surgery
  Recurrence free survival in 3 years
Overall survival in 3 years | Year 3 after surgery
  Overall survival in 3 years

OTHER OUTCOMES:
Quality evaluation index of Lower Mediastinal Lymphadenectomy | through study completion, an average of 3 years
  surgical characteristics that are directly related to the safety outcome of surgery
Learning curve of Lower Mediastinal Lymphadenectomy | through study completion, an average of 3 years
  refers to the number of surgical cases corresponding to the transition point
Treatment tendency of surgeons and patients | through study completion, an average of 3 years
  the proportion of persons willing to receive treatment in randomization
Number of patients that can be screened and successfully recruited | through study completion, an average of 3 years
  The number of patients that can be screened, excluded, successfully recruited, intervented, and followed up throughout each phase of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after the publication of the results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the publication.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Markar SR, Dabakuyo-Yonli TS, Piessen G. Hybrid Minimally Invasive Esophagectomy for Esophageal Cancer. Reply. N Engl J Med. 2019 Apr 25;380(17):e28. doi: 10.1056/NEJMc1901650. No abstract available. PMID 31018084
- [Background] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- [Background] Kurokawa Y, Takeuchi H, Doki Y, Mine S, Terashima M, Yasuda T, Yoshida K, Daiko H, Sakuramoto S, Yoshikawa T, Kunisaki C, Seto Y, Tamura S, Shimokawa T, Sano T, Kitagawa Y. Mapping of Lymph Node Metastasis From Esophagogastric Junction Tumors: A Prospective Nationwide Multicenter Study. Ann Surg. 2021 Jul 1;274(1):120-127. doi: 10.1097/SLA.0000000000003499. PMID 31404008
- [Background] Sugita S, Kinoshita T, Kaito A, Watanabe M, Sunagawa H. Short-term outcomes after laparoscopic versus open transhiatal resection of Siewert type II adenocarcinoma of the esophagogastric junction. Surg Endosc. 2018 Jan;32(1):383-390. doi: 10.1007/s00464-017-5687-6. Epub 2017 Jun 27. PMID 28656339
- [Background] Sugita S, Kinoshita T, Kuwata T, Tokunaga M, Kaito A, Watanabe M, Tonouchi A, Sato R, Nagino M. Long-term oncological outcomes of laparoscopic versus open transhiatal resection for patients with Siewert type II adenocarcinoma of the esophagogastric junction. Surg Endosc. 2021 Jan;35(1):340-348. doi: 10.1007/s00464-020-07406-w. Epub 2020 Feb 5. PMID 32025923
- [Background] Huang CM, Lv CB, Lin JX, Chen QY, Zheng CH, Li P, Xie JW, Wang JB, Lu J, Cao LL, Lin M, Tu RH. Laparoscopic-assisted versus open total gastrectomy for Siewert type II and III esophagogastric junction carcinoma: a propensity score-matched case-control study. Surg Endosc. 2017 Sep;31(9):3495-3503. doi: 10.1007/s00464-016-5375-y. Epub 2016 Dec 15. PMID 27981384
- [Derived] Li S, Ying X, Shan F, Jia Y, Li Z, Xue K, Miao R, Wang Y, Bu Z, Su X, Li Z, Ji J. Laparoscopic vs. open lower mediastinal lymphadenectomy for Siewert type II/III adenocarcinoma of esophagogastric junction: An exploratory, observational, prospective, IDEAL stage 2b cohort study (CLASS-10 study). Chin J Cancer Res. 2022 Aug 30;34(4):406-414. doi: 10.21147/j.issn.1000-9604.2022.04.08. PMID 36199536